CLINICAL TRIAL: NCT04729400
Title: Percutaneous Electrolysis and Vacuum Myofascial Therapy Device in the Treatment of Lateral Epicondylalgia: A Single-Blind Randomized Controlled Trial.
Brief Title: Percutaneous Electrolysis and Vacuum Myofascial Therapy deviceTrial.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Cadiz (Other)
Responsible Party: Principal Investigator, Manuel Rodriguez Huguet, Clinical Professor, University of Cadiz
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Elctrolysis and vacuum
Record Dates: First submitted 2021-01-25; First posted 2021-01-28 (Actual); Last update posted 2022-02-25 (Actual); Status verified 2022-02

CONDITIONS: Epicondylitis
Keywords: Tendinopathy; Electrolysis; Exercise; Dry needing; massage; cupping; vacuum; negative pressure
MeSH Terms: conditions — Tendinopathy; Motor Activity | interventions — Massage

STUDY DESIGN:
Intervention Model Description: A specialist physician will be diagnosed the epicondylitis
Who Masked: Participant
Masking Description: Outcomes assesor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Therapeutic Percutaneous Electrolysis and Vacuum Myofascial Therapy device once week for four weeks associated with eccentric exercises devices at home.
  Interventions: Device: Vacuum Myofascial Therapy device; Procedure: Therapeutic Percutaneous Electrolysis
- CONTROL GROUP (Experimental): The multimodal physical therapy program includes 10 sessions of ultrasound pulsatil therapy (US) and massage associated with eccentric exercises devices at home.
  Interventions: Other: physical therapy program; Procedure: ultrasound pulsatil therapy (US) and massage

INTERVENTIONS:
Device: Vacuum Myofascial Therapy device — Therapeutic Percutaneous Electrolysis and Vacuum Myofascial Therapy device once week for four weeks associated with eccentric exercises devices at home.
  Arms: Experimental group
Other: physical therapy program — The multimodal physical therapy program includes 10 sessions of ultrasound pulsatil therapy (US) and massage associated with eccentric exercises devices at home.
  Arms: CONTROL GROUP
Procedure: Therapeutic Percutaneous Electrolysis — Therapeutic Percutaneous Electrolysis
  Arms: Experimental group
Procedure: ultrasound pulsatil therapy (US) and massage — ultrasound pulsatil therapy (US) and massage
  Arms: CONTROL GROUP

SUMMARY:
The concept of epicondylitis refers to the manifestation of pain in the area of insertion of the epicondile muscles, and that it is accompanied by limitation functional. A tendinopathy is characterized as a process of degeneration, with fibroblast proliferation and disorganization of the fibers of collagen. This tendon pathology especially affects the epicondyle extensors and especially the first and second radial and short extensor carpal.

DETAILED DESCRIPTION:
Experimental group will be treated Therapeutic Percutaneous Electrolysis and Vacuum Myofascial Therapy device once week for four weeks associated with eccentric exercises devices at home and the control group will be included 10 sessions of ultrasound pulsatil therapy (US) and massage associated with eccentric exercises devices at home.

ELIGIBILITY:
Inclusion Criteria:

* Patients of both sexes, aged between 18 and 60 years, in an active state of pain and with a diagnosis of one month of evolution.

Exclusion Criteria:

* Patients who are pregnant, have pacemakers and those surgically operated patients who have been treated with electrolysis and Vacuum Myofascial Therapy Device a month earlier

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2021-06-10 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2021-10-30 (Actual)

PRIMARY OUTCOMES:
The intensity of pain in epicondylitis | Baseline
  A 10-point Numerical Pain Rating Scale (NPRS; 0: no pain, 10: maximum pain) will be used to assess the patients' current level of elbow pain, and the worst and lowest level of pain experienced in the preceding week in the elbow area.

SECONDARY OUTCOMES:
The intensity of pain in epicondylitis | Four and twelve weeks
  A 10-point Numerical Pain Rating Scale (NPRS; 0: no pain, 10: maximum pain) will be used to assess the patients' current level of elbow pain, and the worst and lowest level of pain experienced in the preceding week in the elbow area.
Active elbow range of motion | Baseline,four and twelve weeks
  Measured by a two branches egoniomter
Pressure pain thresholds in epicondylitis trigger points | Baseline, four and twelve weeks
  Pressure pain thresholds (PPTs) will be measured with a pressure algometer (Baseline)
Questionnaire SF 12 | Baseline,four and twelve weeks
  The multidimensional health related quality of life
Scale PRTEE | Baseline,four weeks and Twelve weeks.
  PRTEE is designed to evaluate pain and disability in subjects with lateral elbow tendinopathy. A 10-point Numerical Pain Rating Scale (NPRS; 0: no pain, 10: maximum pain) will be used to assess the patients' current level of elbow pain, and the worst and lowest level of pain experienced in the preceding week in the elbow area.

CONTACTS AND LOCATIONS:
Overall Officials: manuel Rodríguez Huguet, Physiotherapy, Principal Investigator — University of Cádiz
Locations (1):
- Policlínica Santa María, Cadiz, Cádiz, Spain

REFERENCES:
- [Background] Valera-Garrido F, Minaya-Munoz F, Medina-Mirapeix F. Ultrasound-guided percutaneous needle electrolysis in chronic lateral epicondylitis: short-term and long-term results. Acupunct Med. 2014 Dec;32(6):446-54. doi: 10.1136/acupmed-2014-010619. Epub 2014 Aug 13. PMID 25122629
- [Background] Walz DM, Newman JS, Konin GP, Ross G. Epicondylitis: pathogenesis, imaging, and treatment. Radiographics. 2010 Jan;30(1):167-84. doi: 10.1148/rg.301095078. PMID 20083592
- [Background] Rodriguez-Huguet M, Gongora-Rodriguez J, Lomas-Vega R, Martin-Valero R, Diaz-Fernandez A, Obrero-Gaitan E, Ibanez-Vera AJ, Rodriguez-Almagro D. Percutaneous Electrolysis in the Treatment of Lateral Epicondylalgia: A Single-Blind Randomized Controlled Trial. J Clin Med. 2020 Jul 1;9(7):2068. doi: 10.3390/jcm9072068. PMID 32630241
- [Background] Arias-Buria JL, Truyols-Dominguez S, Valero-Alcaide R, Salom-Moreno J, Atin-Arratibel MA, Fernandez-de-Las-Penas C. Ultrasound-Guided Percutaneous Electrolysis and Eccentric Exercises for Subacromial Pain Syndrome: A Randomized Clinical Trial. Evid Based Complement Alternat Med. 2015;2015:315219. doi: 10.1155/2015/315219. Epub 2015 Nov 15. PMID 26649058
- [Background] Garcia Bermejo P, De La Cruz Torres B, Naranjo Orellana J, Albornoz Cabello M. Autonomic Responses to Ultrasound-Guided Percutaneous Needle Electrolysis: Effect of Needle Puncture or Electrical Current? J Altern Complement Med. 2018 Jan;24(1):69-75. doi: 10.1089/acm.2016.0339. Epub 2017 Jan 30. PMID 28135129
- [Background] Rodriguez-Huguet M, Gongora-Rodriguez J, Rodriguez-Huguet P, Ibanez-Vera AJ, Rodriguez-Almagro D, Martin-Valero R, Diaz-Fernandez A, Lomas-Vega R. Effectiveness of Percutaneous Electrolysis in Supraspinatus Tendinopathy: A Single-Blinded Randomized Controlled Trial. J Clin Med. 2020 Jun 12;9(6):1837. doi: 10.3390/jcm9061837. PMID 32545583
- [Background] Kim S, Lee SH, Kim MR, Kim EJ, Hwang DS, Lee J, Shin JS, Ha IH, Lee YJ. Is cupping therapy effective in patients with neck pain? A systematic review and meta-analysis. BMJ Open. 2018 Nov 5;8(11):e021070. doi: 10.1136/bmjopen-2017-021070. PMID 30397006
- [Background] Kim JI, Lee MS, Lee DH, Boddy K, Ernst E. Cupping for treating pain: a systematic review. Evid Based Complement Alternat Med. 2011;2011:467014. doi: 10.1093/ecam/nep035. Epub 2011 Jun 23. PMID 19423657
- [Background] Leem J. Long-term effect of cupping for chronic neck pain. Integr Med Res. 2014 Dec;3(4):217-219. doi: 10.1016/j.imr.2014.10.001. Epub 2014 Oct 14. No abstract available. PMID 28664101
- [Background] Huber R, Emerich M, Braeunig M. Cupping - is it reproducible? Experiments about factors determining the vacuum. Complement Ther Med. 2011 Apr;19(2):78-83. doi: 10.1016/j.ctim.2010.12.006. Epub 2011 Jan 22. PMID 21549258
- [Background] Lauche R, Cramer H, Hohmann C, Choi KE, Rampp T, Saha FJ, Musial F, Langhorst J, Dobos G. The effect of traditional cupping on pain and mechanical thresholds in patients with chronic nonspecific neck pain: a randomised controlled pilot study. Evid Based Complement Alternat Med. 2012;2012:429718. doi: 10.1155/2012/429718. Epub 2011 Dec 7. PMID 22203873
- [Background] Thong ISK, Jensen MP, Miro J, Tan G. The validity of pain intensity measures: what do the NRS, VAS, VRS, and FPS-R measure? Scand J Pain. 2018 Jan 26;18(1):99-107. doi: 10.1515/sjpain-2018-0012. PMID 29794282
- [Background] Rodriguez-Huguet M, Rodriguez-Huguet P, Lomas-Vega R, Ibanez-Vera AJ, Rodriguez-Almagro D. Vacuum myofascial therapy device for non-specific neck pain. A single blind randomized clinical trial. Complement Ther Med. 2020 Aug;52:102449. doi: 10.1016/j.ctim.2020.102449. Epub 2020 May 30. PMID 32951712
- [Background] Gunduz R, Malas FU, Borman P, Kocaoglu S, Ozcakar L. Physical therapy, corticosteroid injection, and extracorporeal shock wave treatment in lateral epicondylitis. Clinical and ultrasonographical comparison. Clin Rheumatol. 2012 May;31(5):807-12. doi: 10.1007/s10067-012-1939-y. Epub 2012 Jan 27. PMID 22278162
- [Derived] Rodriguez-Huguet M, Rodriguez-Almagro D, Rosety-Rodriguez MA, Vinolo-Gil MJ, Molina-Jimenez J, Gongora-Rodriguez J. Pulsed negative pressure myofascial vacuum therapy and percutaneous electrolysis in the treatment of lateral epicondylalgia: A single-blind randomized controlled trial. J Hand Ther. 2024 Oct-Dec;37(4):644-652. doi: 10.1016/j.jht.2024.02.003. Epub 2024 Mar 6. PMID 38453573